CLINICAL TRIAL: NCT05183620
Title: Feeling Hot 2: Evaluating Nocturnal Erection Detection With Penile Temperature Measurements in the Search of a Modern Erectile Dysfunction Diagnostic Tool
Brief Title: Feeling Hot 2: Penile Skin Temperature Measurements of Nocturnal Erections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Hille Torenvlied, Coordinating Investigator, St. Antonius Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 79969
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; RigiScan; Nocturnal erection; Penile temperature
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nocturnal erection measurement (Other): Overnight measurements of the temperature of the penile skin and outer thigh will be performed, while simultaneously the penile circumference and rigidity is determined by RigiScan measurements
  Interventions: Device: Feeling Hot sensor system

INTERVENTIONS:
Device: Feeling Hot sensor system — The Feeling Hot sensor system consists of two temperature probes placed on the penis and the outer thigh of the test subject to measure skin temperature during erection

SUMMARY:
The Feeling Hot studies focus on the proof-of-principle of using temperature sensing as a tool to detect nocturnal erections. In the Feeling Hot 2 study the penile skin temperature is investigated during nocturnal erections during overnight ambulatory measurements. Simultaneous measurements with the RigiScan will be performed to detect the nocturnal erections and validate the principle of temperature measurements for erectile dysfunction diagnostics.

DETAILED DESCRIPTION:
Differentiation in nature of erectile dysfunction (ED) is currently made by nocturnal erection detection with the RigiScan. The RigiScan uses outdated software, measurements are user unfriendly and system components are out of stock. In the search of modernizing erectile dysfunction diagnostics, the question has arisen whether temperature measurements can function as a tool for nocturnal erection detection. With the absence of a pressure component, the patient experience should improve. Literature and mathematical modelling studies have shown that the penile temperature increases significantly during erection. However, no studies have used penile skin temperature measurements to detect nocturnal erections. The Feeling Hot 2 study explores the validity of this measurement set-up for overnight ambulatory measurements of nocturnal erections in the search of modernizing erectile dysfunction diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer without (a history of) erectile dysfunction
* Male
* Aged 18 - 29 years

Exclusion Criteria:

* Test subjects who are unwilling to sign informed consent
* Test subjects with erectile dysfunction
* IIEF-5 score of below 17
* (History of) sickle cell aneamia, atherosclerosis and diabetes type I or II.
* (History of) REM-sleep behavior disorder or other sleep disorders such as restless legs syndrome, insomnia, and sleep apnea
* Usage of sleeping pills or benzodiazepines.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Temperature increase | 8 hours
  Increase in penile skin temperature during nocturnal erection
(De)tumescence duration | 8 hours
  Duration of increased penile skin temperature during erection

SECONDARY OUTCOMES:
Difference between sexual and nocturnal erections | 8 hours
  Penile and outer thigh temperature increase difference between sexual and nocturnal erection

CONTACTS AND LOCATIONS:
Overall Officials: Jack Beck, Dr.,MD., Principal Investigator — Urologist, St. Antonius Ziekenhuis
Locations (1):
- Hille Torenvlied, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No